CLINICAL TRIAL: NCT02765295
Title: Efficacy and Safety of Hydrogen Inhalation on Bronchiectasis (HYBRID): A Randomized, Multi-center, Double-blind, Parallel-group Study
Brief Title: Efficacy and Safety of Hydrogen Inhalation on Bronchiectasis: A Randomized, Multi-center, Double-blind Study
Acronym: HYBRID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Weijie Guan, doctor, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GWJ-2015-H2
Record Dates: First submitted 2016-05-03; First posted 2016-05-06 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Bronchiectasis; Acute Exacerbation of Bronchiectasis; Oxidative Stress
Keywords: Hydrogen; Inhalation; bronchiectasis
MeSH Terms: conditions — Bronchiectasis; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hydrogen inhalation (Active Comparator): The medical ultrasonic nebulizers with hydrogen/oxygen generating function (MUNHO) will be provided exclusively by the sponsor, Asclepius Meditec Inc (Shanghai, China). The MUNHO consists of a electrolytic tank which, by using direct current converted from alternating current (220 V), generates the hydrogen and oxygen gas from pure water (2:1 in volume). The MUNHO is also capable of nebulizing the water via ultrasounds with the hydrogen-oxygen mixture gas which is finally delivered to the patient's airways via the facial mask through a plastic tube. Typically, the volume of hydrogen-oxygen mixed gas is 3 liters per minute (3 L/min). Usual care referred to mucolytics (see below for details) alone or plus chest physiotherapy.
  Interventions: Device: medical ultrasonic hydrogen/oxygen nebulizer (MUNHO)
- oxygen inhalation (Sham Comparator): Oxygen will be generated by an instrument provided by the sponsor, that would be capable of generating oxygen equivalent to that generated by the MUNHO (3L/min mixed gas containing 33.3% oxygen). Usual care referred to mucolytics [[ambroxool (30mg thrice daily), or N-acetylcysteine (0.2g thrice daily)/ serrapeptase (10mg thrice daily), or carbocisteine (500mg thrice daily)] alone or in combination with chest physiotherapy.
  Interventions: Device: Medical molecular mesh oxygen generator

INTERVENTIONS:
Device: medical ultrasonic hydrogen/oxygen nebulizer (MUNHO) — The medical ultrasonic nebulizers with hydrogen/oxygen generating function (MUNHO) will be provided exclusively by the sponsor, Asclepius Meditec Inc (Shanghai, China). The MUNHO consists of a electrolytic tank which, by using direct current converted from alternating current (220 V), generates the hydrogen and oxygen gas from pure water (2:1 in volume). The MUNHO is also capable of nebulizing the water via ultrasounds with the hydrogen-oxygen mixed gas which is finally delivered to the patient's airways via the facial mask through a plastic tube. Typically, the volume of hydrogen-oxygen mixed gas is 3 liters per minute (3 L/min).
  Other Names: hydrogen generating instrument
  Arms: hydrogen inhalation
Device: Medical molecular mesh oxygen generator — medical molecular mesh oxygen generator, type: OLO-1, oxygen flow: 3L/min; Shanghai Ouliang Medical Instrument Inc., Shanghai, China; Registration No.: Shanghai Medical Instrument approval No. 20152540046.
  This device has an identical appearance as compared with the MUHNO so that the patients could not readily discriminate with the MUHNO, and is also capable of displaying the actual cumulative duration of oxygen inhalation.
  Other Names: Oxygen generating instrument
  Arms: oxygen inhalation

SUMMARY:
This is a multi-center, randomized, double-blind, parallel-group trial. After a 2-week run-in period, eligible patients will be, based on the randomization codes kept in sealed envelopes, randomly assigned to receive usual care (mucolytics and/or chest physiotherapy) plus oxygen inahaltion (1 hr daily for 12 consecutive months) or hydrogen inhalation (1 hr daily for 12 consecutive months) provided by the sponsor. At 3 months after the end-of-treatment, a follow-up visit will be scheduled for all patients.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, parallel-group trial. After 2-week run-in period, eligible patients will be, based on the randomization codes kept in sealed envelopes, randomly assigned to two groups.On the basis of usual care [ambroxool (30mg thrice daily), or N-acetylcysteine (0.2g thrice daily)/ serrapeptase (10mg thrice daily), or carbocisteine (500mg thrice daily) and/or chest physiotherapy (10 min, twice daily)], patients were randomized to receive either hydrogen (66.7%, 3L/min, 1 hr twice daily) inhalation or oxygen inhalation (3L/min, 1 hr twice daily) via nasal canula for 12 months. A follow-up visit at month 3 following end-of-treatment was also scheduled. The primary endpoint was the annual frequency of bronchiectasis exacerbations. Hospital visits were scheduled at baseline and months 1, 3, 6, 9, 12 and 15, respectively. At 3 months after the end-of-treatment, a follow-up visit will be scheduled for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients of either gender, ex- or never-smokers, aged between 18 and 75 years
* Clinically stable bronchiectasis, defined as respiratory symptoms and lung function parameters not exceeding normal daily variations and no acute upper respiratory tract infections for 4 consecutive weeks
* Patients with a history of 2 or more bronchiectasis exacerbations (BEs) within the previous 2 years

Exclusion Criteria:

* Other unstable concomitant systemic illnesses (i.e. coronary heart disease, recent cerebral stroke, severe uncontrolled hypertension, active gastric or duodenal ulcer, uncontrolled diabetes, malignancy, hepatic or renal dysfunction)
* Concomitant asthma, allergic bronchopulmonary aspergillosis, or active tuberculosis
* Concomitant chronic obstructive pulmonary disease as the predominant diagnosis
* Treatment with inhaled, oral or systemic antibiotics within 4 weeks
* Type 2 respiratory failure needing oxygen therapy or non-invasive mechanical ventilation
* Females during lactation or pregnancy
* Poor understanding or failure to properly operate the instrument
* Participation in other clinical trials within 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of bronchiectasis exacerbations (BEs) within 12 months | up to 12 months (1 year)
  Frequency of bronchiectasis exacerbations (BEs) within 12 months

SECONDARY OUTCOMES:
Changes in sputum oxidant (hydrogen peroxide, reactive oxygen species) levels at month 6 and 12 as compared with baseline | baseline, month 6 and month 12
  Changes in sputum oxidant (hydrogen peroxide, reactive oxygen species) levels at month 6 and 12 as compared with baseline
Time to the first bronchiectasis exacerbations (BEs) within 12 months | up to 12 months
  Time to the first bronchiectasis exacerbations (BEs) within 12 months
Changes in sputum antioxidants levels (catalase, superoxide dismutase and total antioxidant capacity) at month 6 and 12 as compared with baseline | baseline, month 6 and month 12
  Changes in sputum antioxidants levels (catalase, superoxide dismutase and total antioxidant capacity) at month 6 and 12 as compared with baseline
Changes in serum oxidant (hydrogen peroxide, reactive oxygen species) levels at month 6 and 12 as compared with baseline | baseline, month 6 and month 12
  Changes in serum oxidant (hydrogen peroxide, reactive oxygen species) levels at month 6 and 12 as compared with baseline
Changes in serum antioxidants levels (catalase, superoxide dismutase and total antioxidant capacity) at month 6 and 12 as compared with baseline | baseline, month 6 and month 12
  Changes in serum antioxidants levels (catalase, superoxide dismutase and total antioxidant capacity) at month 6 and 12 as compared with baseline
Changes in spirometry, including FEV1, FEV1/FVC ratio and MMEF at each visit following randomization as compared with baseline | baseline, month 1, month 3, month 6, month 9 and month 12
  Changes in spirometry, including FEV1, FEV1/FVC ratio and MMEF at each visit following randomization as compared with baseline
Changes in CRP levels at month 6 and 12 as compared with baseline | baseline, month 6 and month 12
  Changes in CRP levels at month 6 and 12 as compared with baseline
Changes in quality of life assessed by using Quality-of-Life Questionnaire--Bronchiectasis (QoL-B) at month 6 and 12 as compared with baseline | baseline, month 6 and month 12
  Changes in quality of life assessed by using Quality-of-Life Questionnaire--Bronchiectasis (QoL-B) at month 6 and 12 as compared with baseline

OTHER OUTCOMES:
Changes in airway impedance as measured by impulse oscillometry (Z5, R5, R20, X5, Fres and AX at each visit as compared with baseline | baseline, month 1, month 3, month 6, month 9 and month 12
  Changes in airway impedance as measured by impulse oscillometry (Z5, R5, R20, X5, Fres and AX at each visit as compared with baseline
Changes in dyshomogeneity (lung clearance index) at month 6 and 12 as compared with baseline | baseline, month 6 and month 12
  Changes in dyshomogeneity (lung clearance index) at month 6 and 12 as compared with baseline
Changes in anaerobic threshold (during cardiopulmonary exercise testing) at month 6 and 12 as compared with baseline | baseline, month 6 and month 12
  Changes in anaerobic threshold (during cardiopulmonary exercise testing) at month 6 and 12 as compared with baseline
Changes in oxygen pulse (during cardiopulmonary exercise testing) at month 6 and 12 as compared with baseline | baseline, month 6 and month 12
  Changes in oxygen pulse (during cardiopulmonary exercise testing) at month 6 and 12 as compared with baseline
Changes in the difference of arterial and alveolar oxygen partial pressure (during cardiopulmonary exercise testing) at month 6 and 12 as compared with baseline | baseline, month 6 and month 12
  Changes in the difference of arterial and alveolar oxygen partial pressure (during cardiopulmonary exercise testing) at month 6 and 12 as compared with baseline
Changes in carbon dioxide ventilatory equivalent (during cardiopulmonary exercise testing) at month 6 and 12 as compared with baseline | baseline, month 6 and month 12
  Changes in carbon dioxide ventilatory equivalent (during cardiopulmonary exercise testing) at month 6 and 12 as compared with baseline
Changes in 24-hour sputum volume at each visit as compared with baseline | baseline, month 1, month 3, month 6, month 9 and month 12
  Changes in 24-hour sputum volume at each visit as compared with baseline
Changes in the levels of sputum inflammatory markers (interleukin-6, interleukin-8 and tumor necrosis factor-α) at month 6 and 12 as compared with baseline | baseline, month 6 and month 12
  Changes in the levels of sputum inflammatory markers (interleukin-6, interleukin-8 and tumor necrosis factor-α) at month 6 and 12 as compared with baseline
Changes in sputum matrix metalloproteinases (MMP-8, MMP-9, MMP-9/TIMP-1 ratio) levels at month 6 and 12 as compared with baseline | baseline, month 6 and month 12
  Changes in sputum matrix metalloproteinases (MMP-8, MMP-9, MMP-9/TIMP-1 ratio) levels at month 6 and 12 as compared with baseline
The rates of Pseudomonas aeruginosa isolated from sputum at baseline and end-of-treatment at month 6 and 12 as compared with baseline | baseline, month 6 and month 12
  The rates of Pseudomonas aeruginosa isolated from sputum at baseline and end-of-treatment at month 6 and 12 as compared with baseline
Sputum microbiota compositions before and after hydrogen therapy | up to 12 months (at baseline, month 6, and month 12)
  Sputum microbiota compositions before and after hydrogen therapy. This is an exploratory outcome.
the rate of adverse events | up to 12 months
  the rate of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Nan-shan Zhong, MD, Study Chair — Guangzhou Institute of Respiratory Disease
Locations (5):
- China (5):
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - West China Hospital Affiliateyd to Sichuan Universit, Chengdu
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pasteur MC, Bilton D, Hill AT; British Thoracic Society Bronchiectasis non-CF Guideline Group. British Thoracic Society guideline for non-CF bronchiectasis. Thorax. 2010 Jul;65 Suppl 1:i1-58. doi: 10.1136/thx.2010.136119. PMID 20627931
- [Background] Loebinger MR, Wells AU, Hansell DM, Chinyanganya N, Devaraj A, Meister M, Wilson R. Mortality in bronchiectasis: a long-term study assessing the factors influencing survival. Eur Respir J. 2009 Oct;34(4):843-9. doi: 10.1183/09031936.00003709. Epub 2009 Apr 8. PMID 19357155
- [Background] Barker AF. Bronchiectasis. N Engl J Med. 2002 May 2;346(18):1383-93. doi: 10.1056/NEJMra012519. No abstract available. PMID 11986413
- [Background] Loukides S, Horvath I, Wodehouse T, Cole PJ, Barnes PJ. Elevated levels of expired breath hydrogen peroxide in bronchiectasis. Am J Respir Crit Care Med. 1998 Sep;158(3):991-4. doi: 10.1164/ajrccm.158.3.9710031. PMID 9731036
- [Background] Horvath I, Loukides S, Wodehouse T, Kharitonov SA, Cole PJ, Barnes PJ. Increased levels of exhaled carbon monoxide in bronchiectasis: a new marker of oxidative stress. Thorax. 1998 Oct;53(10):867-70. doi: 10.1136/thx.53.10.867. PMID 10193374
- [Background] Wood LG, Garg ML, Simpson JL, Mori TA, Croft KD, Wark PA, Gibson PG. Induced sputum 8-isoprostane concentrations in inflammatory airway diseases. Am J Respir Crit Care Med. 2005 Mar 1;171(5):426-30. doi: 10.1164/rccm.200408-1010OC. Epub 2004 Dec 3. PMID 15579724
- [Background] Olveira G, Olveira C, Dorado A, Garcia-Fuentes E, Rubio E, Tinahones F, Soriguer F, Murri M. Cellular and plasma oxidative stress biomarkers are raised in adults with bronchiectasis. Clin Nutr. 2013 Feb;32(1):112-7. doi: 10.1016/j.clnu.2012.06.002. Epub 2012 Jun 29. PMID 22749311
- [Background] Ohsawa I, Ishikawa M, Takahashi K, Watanabe M, Nishimaki K, Yamagata K, Katsura K, Katayama Y, Asoh S, Ohta S. Hydrogen acts as a therapeutic antioxidant by selectively reducing cytotoxic oxygen radicals. Nat Med. 2007 Jun;13(6):688-94. doi: 10.1038/nm1577. Epub 2007 May 7. PMID 17486089
- [Background] Sun Q, Cai J, Liu S, Liu Y, Xu W, Tao H, Sun X. Hydrogen-rich saline provides protection against hyperoxic lung injury. J Surg Res. 2011 Jan;165(1):e43-9. doi: 10.1016/j.jss.2010.09.024. Epub 2010 Oct 15. PMID 21067781
- [Background] Huang CS, Kawamura T, Peng X, Tochigi N, Shigemura N, Billiar TR, Nakao A, Toyoda Y. Hydrogen inhalation reduced epithelial apoptosis in ventilator-induced lung injury via a mechanism involving nuclear factor-kappa B activation. Biochem Biophys Res Commun. 2011 May 6;408(2):253-8. doi: 10.1016/j.bbrc.2011.04.008. Epub 2011 Apr 5. PMID 21473852
- [Background] Kawamura T, Wakabayashi N, Shigemura N, Huang CS, Masutani K, Tanaka Y, Noda K, Peng X, Takahashi T, Billiar TR, Okumura M, Toyoda Y, Kensler TW, Nakao A. Hydrogen gas reduces hyperoxic lung injury via the Nrf2 pathway in vivo. Am J Physiol Lung Cell Mol Physiol. 2013 May 15;304(10):L646-56. doi: 10.1152/ajplung.00164.2012. Epub 2013 Mar 8. PMID 23475767
- [Background] Terasaki Y, Ohsawa I, Terasaki M, Takahashi M, Kunugi S, Dedong K, Urushiyama H, Amenomori S, Kaneko-Togashi M, Kuwahara N, Ishikawa A, Kamimura N, Ohta S, Fukuda Y. Hydrogen therapy attenuates irradiation-induced lung damage by reducing oxidative stress. Am J Physiol Lung Cell Mol Physiol. 2011 Oct;301(4):L415-26. doi: 10.1152/ajplung.00008.2011. Epub 2011 Jul 15. PMID 21764987
- [Background] Zheng J, Liu K, Kang Z, Cai J, Liu W, Xu W, Li R, Tao H, Zhang JH, Sun X. Saturated hydrogen saline protects the lung against oxygen toxicity. Undersea Hyperb Med. 2010 May-Jun;37(3):185-92. PMID 20568549
- [Background] Ning Y, Shang Y, Huang H, Zhang J, Dong Y, Xu W, Li Q. Attenuation of cigarette smoke-induced airway mucus production by hydrogen-rich saline in rats. PLoS One. 2013 Dec 20;8(12):e83429. doi: 10.1371/journal.pone.0083429. eCollection 2013. PMID 24376700
- [Background] Xiao M, Zhu T, Wang T, Wen FQ. Hydrogen-rich saline reduces airway remodeling via inactivation of NF-kappaB in a murine model of asthma. Eur Rev Med Pharmacol Sci. 2013 Apr;17(8):1033-43. PMID 23661516
- [Background] Kajiyama S, Hasegawa G, Asano M, Hosoda H, Fukui M, Nakamura N, Kitawaki J, Imai S, Nakano K, Ohta M, Adachi T, Obayashi H, Yoshikawa T. Supplementation of hydrogen-rich water improves lipid and glucose metabolism in patients with type 2 diabetes or impaired glucose tolerance. Nutr Res. 2008 Mar;28(3):137-43. doi: 10.1016/j.nutres.2008.01.008. PMID 19083400
- [Background] Nakao A, Toyoda Y, Sharma P, Evans M, Guthrie N. Effectiveness of hydrogen rich water on antioxidant status of subjects with potential metabolic syndrome-an open label pilot study. J Clin Biochem Nutr. 2010 Mar;46(2):140-9. doi: 10.3164/jcbn.09-100. Epub 2010 Feb 24. PMID 20216947
- [Background] Kang KM, Kang YN, Choi IB, Gu Y, Kawamura T, Toyoda Y, Nakao A. Effects of drinking hydrogen-rich water on the quality of life of patients treated with radiotherapy for liver tumors. Med Gas Res. 2011 Jun 7;1(1):11. doi: 10.1186/2045-9912-1-11. PMID 22146004
- [Background] Ishibashi T, Sato B, Rikitake M, Seo T, Kurokawa R, Hara Y, Naritomi Y, Hara H, Nagao T. Consumption of water containing a high concentration of molecular hydrogen reduces oxidative stress and disease activity in patients with rheumatoid arthritis: an open-label pilot study. Med Gas Res. 2012 Oct 2;2(1):27. doi: 10.1186/2045-9912-2-27. PMID 23031079
- [Background] Ishibashi T, Sato B, Shibata S, Sakai T, Hara Y, Naritomi Y, Koyanagi S, Hara H, Nagao T. Therapeutic efficacy of infused molecular hydrogen in saline on rheumatoid arthritis: a randomized, double-blind, placebo-controlled pilot study. Int Immunopharmacol. 2014 Aug;21(2):468-73. doi: 10.1016/j.intimp.2014.06.001. Epub 2014 Jun 11. PMID 24929023
- [Background] Guan WJ, Gao YH, Xu G, Lin ZY, Tang Y, Li HM, Lin ZM, Zheng JP, Chen RC, Zhong NS. Capsaicin cough sensitivity and the association with clinical parameters in bronchiectasis. PLoS One. 2014 Nov 19;9(11):e113057. doi: 10.1371/journal.pone.0113057. eCollection 2014. PMID 25409316
- [Background] Guan WJ, Gao YH, Xu G, Lin ZY, Tang Y, Li HM, Lin ZM, Zheng JP, Chen RC, Zhong NS. Characterization of lung function impairment in adults with bronchiectasis. PLoS One. 2014 Nov 18;9(11):e113373. doi: 10.1371/journal.pone.0113373. eCollection 2014. PMID 25405614
- [Background] Gao Y, Guan W, Xu G, Lin Z, Tang Y, Lin Z, Li H, Gao Y, Luo Q, Zhong N, Chen R. Sleep disturbances and health-related quality of life in adults with steady-state bronchiectasis. PLoS One. 2014 Jul 18;9(7):e102970. doi: 10.1371/journal.pone.0102970. eCollection 2014. PMID 25036723
- [Background] Gao YH, Guan WJ, Xu G, Gao Y, Lin ZY, Tang Y, Lin ZM, Li HM, Luo Q, Zhong NS, Birring SS, Chen RC. Validation of the Mandarin Chinese version of the Leicester Cough Questionnaire in bronchiectasis. Int J Tuberc Lung Dis. 2014 Dec;18(12):1431-7. doi: 10.5588/ijtld.14.0195. PMID 25517807
- [Background] Gao YH, Guan WJ, Xu G, Lin ZY, Tang Y, Lin ZM, Gao Y, Li HM, Zhong NS, Zhang GJ, Chen RC. The role of viral infection in pulmonary exacerbations of bronchiectasis in adults: a prospective study. Chest. 2015 Jun;147(6):1635-1643. doi: 10.1378/chest.14-1961. PMID 25412225
- [Background] Guan WJ, Gao YH, Xu G, Lin ZY, Tang Y, Li HM, Lin ZM, Zheng JP, Chen RC, Zhong NS. Six-minute walk test in Chinese adults with clinically stable bronchiectasis: association with clinical indices and determinants. Curr Med Res Opin. 2015 Apr;31(4):843-52. doi: 10.1185/03007995.2015.1013625. Epub 2015 Mar 3. PMID 25708564
- [Background] Guan WJ, Gao YH, Xu G, Lin ZY, Tang Y, Li HM, Lin ZM, Zheng JP, Chen RC, Zhong NS. Impulse oscillometry in adults with bronchiectasis. Ann Am Thorac Soc. 2015 May;12(5):657-65. doi: 10.1513/AnnalsATS.201406-280OC. PMID 25654540
- [Background] Guan WJ, Gao YH, Xu G, Lin ZY, Tang Y, Li HM, Lin ZM, Zheng JP, Chen RC, Zhong NS. Aetiology of bronchiectasis in Guangzhou, southern China. Respirology. 2015 Jul;20(5):739-48. doi: 10.1111/resp.12528. Epub 2015 Mar 26. PMID 25819403
- [Background] Guan WJ, Gao YH, Xu G, Lin ZY, Tang Y, Li HM, Lin ZM, Zheng JP, Chen RC, Zhong NS. Sputum bacteriology in steady-state bronchiectasis in Guangzhou, China. Int J Tuberc Lung Dis. 2015 May;19(5):610-9. doi: 10.5588/ijtld.14.0613. PMID 25868032
- [Background] Tsang KW, Chan K, Ho P, Zheng L, Ooi GC, Ho JC, Lam W. Sputum elastase in steady-state bronchiectasis. Chest. 2000 Feb;117(2):420-6. doi: 10.1378/chest.117.2.420. PMID 10669685
- [Background] Tsang KW, Ho PL, Lam WK, Ip MS, Chan KN, Ho CS, Ooi CC, Yuen KY. Inhaled fluticasone reduces sputum inflammatory indices in severe bronchiectasis. Am J Respir Crit Care Med. 1998 Sep;158(3):723-7. doi: 10.1164/ajrccm.158.3.9710090. PMID 9730996
- [Background] Chalmers JD, Goeminne P, Aliberti S, McDonnell MJ, Lonni S, Davidson J, Poppelwell L, Salih W, Pesci A, Dupont LJ, Fardon TC, De Soyza A, Hill AT. The bronchiectasis severity index. An international derivation and validation study. Am J Respir Crit Care Med. 2014 Mar 1;189(5):576-85. doi: 10.1164/rccm.201309-1575OC. PMID 24328736
- [Background] Rowan SA, Bradley JM, Bradbury I, Lawson J, Lynch T, Gustafsson P, Horsley A, O'Neill K, Ennis M, Elborn JS. Lung clearance index is a repeatable and sensitive indicator of radiological changes in bronchiectasis. Am J Respir Crit Care Med. 2014 Mar 1;189(5):586-92. doi: 10.1164/rccm.201310-1747OC. PMID 24428575
- [Background] Horsley AR, Gustafsson PM, Macleod KA, Saunders C, Greening AP, Porteous DJ, Davies JC, Cunningham S, Alton EW, Innes JA. Lung clearance index is a sensitive, repeatable and practical measure of airways disease in adults with cystic fibrosis. Thorax. 2008 Feb;63(2):135-40. doi: 10.1136/thx.2007.082628. Epub 2007 Aug 3. PMID 17675315
- [Background] Quittner AL, O'Donnell AE, Salathe MA, Lewis SA, Li X, Montgomery AB, O'Riordan TG, Barker AF. Quality of Life Questionnaire-Bronchiectasis: final psychometric analyses and determination of minimal important difference scores. Thorax. 2015 Jan;70(1):12-20. doi: 10.1136/thoraxjnl-2014-205918. Epub 2014 Oct 16. PMID 25323621
- [Background] Billinger SA, Vidoni ED, Honea RA, Burns JM. Cardiorespiratory response to exercise testing in individuals with Alzheimer's disease. Arch Phys Med Rehabil. 2011 Dec;92(12):2000-5. doi: 10.1016/j.apmr.2011.07.194. PMID 22133248